CLINICAL TRIAL: NCT00545220
Title: Problem Solving Training and Low Vision Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X060817006; 5K23EY017327-02 (NIH)
Record Dates: First submitted 2007-09-21; First posted 2007-10-17 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): PST
  Interventions: Behavioral: problem-solving training
- 2 (Sham Comparator): Attention Control
  Interventions: Behavioral: sham intervention

INTERVENTIONS:
Behavioral: problem-solving training
  Arms: 1
Behavioral: sham intervention
  Arms: 2

SUMMARY:
Vision loss can result in feelings of frustration, helplessness, anxiety, depression, and anger, which compromise a person's activities of everyday living. While emotional distress may resolve in some persons without intervention, unmanaged and persistent distress places the person at risk for continued decrements in health status and the potential development of more severe conditions (i.e., depression, poor health outcomes). Persons with low vision will be recruited and randomly assigned to either an innovative, problem-solving training (PST) intervention group designed specifically for persons with low vision or a sham intervention/control group. Primary and secondary outcomes will be assessed at baseline prior to intervention and at 3 month follow-up, 7 month follow-up, 12 month follow-up, and 24 month follow-up by a research interviewer masked to participants' randomization. This project will: (1) demonstrate how specified physical and emotional outcomes of persons with low vision change across time, (2) evaluate the effectiveness of a PST intervention that will be delivered to persons with low vision; and (3) identify persons with low vision who are at risk for adverse emotional and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* +19 yrs of age
* Underwent a low vision rehabilitation initial eye exam
* No more than 2 errors on cognitive on cognitive screening measure (SPBS)
* Must have access to telephone
* No significant hearing problems
* No significant communication problems
* Speaks fluent English

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2007-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies Depression Scale (CES-D) | baseline, 3months, 6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dreer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States